CLINICAL TRIAL: NCT04619953
Title: Neuropsychological Changes After Cognitive-motor Dual Task Training in Patients With Multiple Sclerosis
Brief Title: Cognitive-motor Dual Task Training in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, Head of Rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE/PROG.812
Record Dates: First submitted 2020-10-28; First posted 2020-11-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; Cognitive Impairment; Motor Disorders
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Motor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural Stability group (PSg) (Active Comparator): The Postural Stability group (PSg) will perform 30 minutes of conventional neuromotor rehabilitation and 20 minutes of dynamic postural stability training.
  Interventions: Other: Dynamic Postural Stability Training; Other: Conventional Therapy
- Cognitive-Motor group (CMg) (Active Comparator): The Cognitive-Motor group (CMg) performed 30 minutes of conventional neuromotor rehabilitation and 20 minutes of cognitive-motor training.
  Interventions: Other: Cognitive-Motor Training; Other: Conventional Therapy

INTERVENTIONS:
Other: Dynamic Postural Stability Training — The dynamic postural stability training, will consist of marching on unstable surface and on treadmill both with open and with closed eyes.
  Arms: Postural Stability group (PSg)
Other: Cognitive-Motor Training — The cognitive-motor training consisted of a dual task paradigm: each patient was asked to walk without stopping and was explained that, during the task, they might hear a sound, and in that case, they should have look at the stimulus 'side and recognize a visual target. This dual task was performed both marching on an unstable surface and marching on treadmill.
  Arms: Cognitive-Motor group (CMg)
Other: Conventional Therapy — The conventional neuromotor rehabilitation will consist in muscles stretching, active-assisted mobilizations, neuromuscular facilitations, gait training and balance exercises using swinging platforms

SUMMARY:
Clinical features of Multiple Sclerosis (MS) vary widely from patient to other. About the 60% of patients with MS presents cognitive deficits associated with motor disability. The principal consequences of the motor disabilities concern difficult in gait and balance. The principal cognitive deficits concern the speed in elaborating information, the complex attention and the memory. During walking in daily life, it is often required to turn the head for looking something happening in the surrounding environment, for example when a sudden noise is heard, while crossing the street, when there's something interesting around or when is required to verbally answer to someone without stopping walking. All these examples are referred to a common daily life mechanism that has been defined as dual task (DT). Considering that the attention is a limited function, divide it in two different and simultaneous tasks (motor and cognitive), cause a cognitive-motor interference (CMI) that lead to a loss of efficacy in one or in both the tasks. The main aim of the study is to verify the impact of a brief rehabilitation training that combining motor and cognitive therapy using a dual-task paradigm, on balance and gait in MS patients, compared with the traditional therapies that provide a specific postural stability rehabilitation approach. Recruited patients will be randomized in two different groups which perform two different training. Each group perform the allocated training 3 times a week for 4 weeks. All the patients will be evaluated at the baseline (T0), at the end of the training (T1) and 60 days after the end of the training (T2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according with revisited McDonalds criteria;
* Expanded Disability Status Scale (EDSS) ranging between 0 and 6;
* Ability to walk independently or with aid for at least 50 meters.

Exclusion Criteria:

* Associated psychiatric and/or neurological disorders (different from the MS);
* Clinical relapse within the three months prior to enrollment;
* Steroid therapy within 30 days before the enrollment;
* Peripheric diseases as visual and/or auditory impairments that could interfere with motor and cognitive tasks execution;
* Fracture of lower limb within three months before the enrollment.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation System Test (Mini-BESTest) | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of MiniBestTest (MBT) from baseline at 4 weeks of the training and at 60 days after the end of the training. The Mini-BESTest values ranging from 0 to 28, where 0 means the worse outcome and 28 the best one.

SECONDARY OUTCOMES:
Modified Barthel Index (MBI) | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of Modified Barthel Index (MBI) from baseline at 4 weeks of the training and at 60 days after the end of the training. MBI values ranging from 0 to 105, where 0 means the worse outcome and 105 the best one
Tinetti Balance and Gait Scale (TBG) | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of Tinetti Balance and Gait Scale (TBG) from baseline at 4 weeks of the training and at 60 days after the end of the training. TBG values ranging from 0 to 28, where 0 means the worse outcome and 28 the best one
10 Meter Walk Test (10MWT) | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of 10 Meter Walk Test (10MWT) from baseline at 4 weeks of the training and at 60 days after the end of the training. 10MWT allows to evaluate the walking speed.
Inertial sensors-based assessment | Baseline, after 4 weeks of training, and 2 months after the end of training
  Set of seven magneto-inertial sensors (Opal, APDM Inc., Portland, Oregon, USA) will be used during the execution of walking motor tasks.
  Changes of continuous accelerometer signals will be recorded from baseline at 4 weeks of the training and at 60 days after the end of the training
2 Minute Walking Test (2MWT) | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of 2 Minute Walking Test (2MWT) from baseline at 4 weeks of the training and at 60 days after the end of the training. 2MWT allows to evaluate the endurance assessing the walking distance over two minutes
2 Minute Walking Test (2MWT) associated with Cognitive Task | Baseline, after 4 weeks of training, and 2 months after the end of training
  Change of 2 Minute Walking Test (2MWT) associated with Cognitive Task from baseline at 4 weeks of the training and at 60 days after the end of the training. 2MWT associated with Cognitive Task allows to evaluate the endurance assessing the walking distance over two minutes during a cognitive task execution (ex: verbalize the the highest number of animals'names during walking)

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tramontano, Roma, Italy